CLINICAL TRIAL: NCT02479217
Title: Safety of Xeloda in Solid Tumours
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20367
Record Dates: First submitted 2015-05-27; First posted 2015-06-24 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer, Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Adjuvant therapy: Patients prescribed Xeloda per registered indicatilons were observed until disease progression or 8 cycles for adjuvant colon cancer
  Interventions: Drug: Xeloda
- Combination Therapy: Patients prescribed Xeloda with docetaxel for metastatic breast cancer after failure to anthacyclines were observed until disease progression
  Interventions: Drug: Docetaxel; Drug: Xeloda
- Monotherapy: Patients prescribed Xeloda per registered indicatilons were observed until disease progression or 8 cycles for adjuvant colon cancer
  Interventions: Drug: Xeloda

INTERVENTIONS:
Drug: Docetaxel
  Groups: Combination Therapy
Drug: Xeloda

SUMMARY:
The primary objective of this study is to observe safety and tolerability of Xeloda as used in medical practice, alone and in combination with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

Metastatic Breast Cancer:

* women >=18 years of age
* Patients with locally advanced or metastatic breast cancer after failure of cytotoxic chemotherapy.
* Previous therapy should have included an anthracycline.
* Patients with locally advanced or metastatic breast cancer after failure of taxanes and an anthracycline-containing chemotherapy regimen or for whom further anthracycline therapy is not indicated.
* Female patients with histopathologically proven metastatic breast cancer
* Adequate bone marrow, liver, renal and cardiac functions

Colon Cancer:

* Patients >18 years of age
* Patients with histologicaly confirmed colon cancer
* Patients with potential curative tumor resection within 8 weeks before enrolment in the study
* Patients previously not treated with chemiotherapy

Exclusion Criteria:

Metastatic Breast Cancer:

* Patients previously treated with docetaxel (Taxotere) or capecitabine (Xeloda)
* Patients with contraindications for any of study drugs as listed in approved SmPC

Colon Cancer:

* Patients previously treated with chemiotherapy
* Patients with contraindications for study drug as listed in approved SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early or metastatic colon cancer, and patients with metastatic breast cancer, no age limit
Sampling Method: Non-Probability Sample
Enrollment: 1268 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | within 18 months

SECONDARY OUTCOMES:
Disease free survival (DFS) | within 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Kamenitz, Serbia